CLINICAL TRIAL: NCT03266614
Title: "Recovery 4 US" - A Photovoice-based Social Media Program to Enhance the Recovery and Community Participation of Individuals With Psychiatric Disabilities
Brief Title: "Recovery 4 US" - A Photovoice-based Social Media Program
Acronym: R4US
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Responsible Party: Principal Investigator, Zlatka Russinova, Research Associate Professor, Boston University Charles River Campus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 4458
Record Dates: First submitted 2017-08-28; First posted 2017-08-30 (Actual); Last update posted 2018-11-30 (Actual); Status verified 2018-11

CONDITIONS: Mental Illness; Social Isolation; Loneliness
Keywords: Mental Illness; Loneliness; Hope; Community; Social Media
MeSH Terms: conditions — Mental Disorders; Social Isolation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Recovery 4 US (Experimental): This group receives a smartphone with the Recovery 4 US application and access to the application website.
  Interventions: Behavioral: Recovery 4 Us
- Services as usual (No Intervention): This group receives a smartphone but no access to the Recovery 4 US application.

INTERVENTIONS:
Behavioral: Recovery 4 Us — R4US is a social media program aimed at the enhancement of community participation and overall recovery of individuals with psychiatric disabilities.
  Other Names: R4US
  Arms: Recovery 4 US

SUMMARY:
This study is a randomized trial evaluating "Recovery 4 US", a social media program aimed at the enhancement of community participation and overall recovery of individuals with psychiatric disabilities.This innovative e-mental health program integrates Internet and mobile technologies and is designed to be a self-sustaining recovery-oriented virtual community for individuals living with a disabling mental illness based on the principles of Photovoice.

DETAILED DESCRIPTION:
This study is a randomized trial evaluating "Recovery 4 US", a social media program aimed at the enhancement of community participation and overall recovery of individuals with psychiatric disabilities.This innovative e-mental health program integrates Internet and mobile technologies and is designed to be a self-sustaining recovery-oriented virtual community for individuals living with a disabling mental illness based on the principles of Photovoice.

The "Recovery 4 US" program which includes a mobile phone application and a password protected website, has three main components: 1) receipt of daily hope-inspiring message, paired with a corresponding visual image; 2) creation and viewing of recovery-oriented Photovoice works; and 3) opportunity to attend community events initiated by members of the "Recovery 4 US" community.

The benefits of the "Recovery 4 US" program will be evaluated through a randomized trial with n=60 participants. The study will take place at the Boston University Center for Psychiatric Rehabilitation. Participants will be randomized to the experimental group (provided with a smartphone and access to "Recovery 4 US" application and website) or the control group (provided with a smartphone but without access to the "Recovery 4 US" app or website). We anticipate participation in the program will be associated with reduced loneliness, increased hopefulness, community participation, and overall recovery.

The recruitment goal for this study was amended to n=70.

ELIGIBILITY:
Inclusion Criteria:

* are 18 or older
* have been recipients of services at the BU CPR Recovery Center due to having a DSM-V diagnosis of mental illness, including dual diagnosis (dual diagnosis refers to co-occurring mental illness and alcohol/ substance use disorder) as indicated in their records
* are interested in participating in a social media program
* are fluent in English
* have a basic ability to use a mobile phone

Exclusion Criteria:

* Inability to give full and knowing consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2017-04-07 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
UCLA Loneliness Scale | Change from Baseline to 3 months to 6 months
  A 20-item 4-point Likert-type scale, widely used measure of loneliness and social isolation with Cronbach's alpha coefficients ranging from .89 to .94

SECONDARY OUTCOMES:
Herth Hope Index | Change from Baseline to 3 months to 6 months
  12 item 4-point Likert type scale measuring the level of generalized hopefulness of the individual; the reported Cronbach's alpha coefficient of internal consistency of the scale is .97
Perceived Stress Scale | Change from Baseline to 3 months to 6 months
  10-item 5-point Likert-type scale self-report measure of the level of stress experienced at a given point of time. It was designed to capture how unpredictable, uncontrollable and overloaded respondents find their lives based on their capacity to cope with stress. Reported internal consistency coefficients for the scale ranged between 0.90 and 0.92
Multi-Dimensional Assessment of Community Participation | Change from Baseline to 3 months to 6 months
  Consists of objective and subjective measures of community belonging, inclusion and participation
Recovery Assessment Scale | Change from Baseline to 3 months to 6 months
  24-item 5-point Likert rating scale assessing the level of overall recovery among people with psychiatric disabilities.
BASIS-R | Change from Baseline to 3 months to 6 months
  measures: mood disturbances, anxiety, interpersonal and role functioning, daily living skills, psychotic symptoms, impulsivity and substance use on a scale from no difficulty to extreme difficulty.

CONTACTS AND LOCATIONS:
Overall Officials: Zlatka Russinova, PhD, Principal Investigator — Boston University
Locations (1):
- Boston University Center for Psychiatric Rehabilitation, Boston, Massachusetts, United States